CLINICAL TRIAL: NCT05842408
Title: A Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of DA-5212 in Patients with Functional Dyspepsia
Brief Title: Clinical Trial of DA-5212 in Patients with Functional Dyspepsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA5212_FDQ_III
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DA-5212 (Experimental): administered once daily for 4weeks
  Interventions: Drug: DA-5212
- DA-5212-R (Other): administered once daily for 4weeks
  Interventions: Drug: DA-5212-R

INTERVENTIONS:
Drug: DA-5212 — Test drug: DA-5212
  Arms: DA-5212
Drug: DA-5212-R — Control drug: DA-5212-R
  Arms: DA-5212-R

SUMMARY:
This study is to evaluate efficacy and safety of DA-5212 in patients with functional dyspepsia

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 19 years of age
* Patients who diagnosed with functional dyspepsia
* Patients with no organic cause for digestive symptoms found by upper gastrointestinal endoscopy at screening visit

Exclusion Criteria:

* Patients with organic disease or medical history that may cause dyspepsia within 6 months before screening visit
* Patients who have a history of drugs or alcohol abuse and dependence within 6 months before screening visit
* Patients with hypersensitivity to investigational drugs and similar drugs
* Pregnant or breastfeeding women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Change in NDI-K functional dyspepsia score | Change from baseline at 4 weeks

SECONDARY OUTCOMES:
Change in overall treatment score of patients | Change from baseline at 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Wonkwang University Hospital, Iksan, Muwangro 895, South Korea